CLINICAL TRIAL: NCT01017224
Title: DAHANCA 24: Prognostic Value of 18F-FAZA Positron Emission Tomography After Primary Curative Radiotherapy for Squamous Cell Carcinoma of the Head and Neck
Brief Title: DAHANCA 24: Prognostic Value of 18F-FAZA in Head and Neck Squamous Cell Carcinoma (HNSCC)
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Danish Head and Neck Cancer Group (Network)
Responsible Party: Sponsor
Other Study IDs: DAHANCA 24
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Cancer of the Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — fluoroazomycin arabinoside

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: 18F-FAZA — PET scan

SUMMARY:
Solid tumours contain varying degrees of hypoxia. Studies show hypoxia to be associated with poor local control and survival, as hypoxia is a cause of resistance to radio- and chemotherapy and the development of a more aggressive tumour.

Previous attempts to measure hypoxia have been biased because the techniques have been invasive, not repeatable or difficult to apply on a routine basis. There is great interest in trying to measure hypoxia in tumours as this could lead to individualized hypoxia-modifying therapy and prediction of treatment response. Additionally the investigators' knowledge of change in hypoxia over time is limited, but of great interest as individualised treatment, such as intensity-modulated radiation therapy (IMRT) is emerging.

18F-FAZA, appears promising. It is a nitroimidazole, which gets trapped in hypoxic cells and can be detected by a positron emission therapy (PET) scan. Compared to other nitroimidazoles, 18F-FAZA has superior biokinetics and thereby is believed to provide a faster and clearer image of hypoxia.

The investigators' hypothesis is that 18F-FAZA can be used as a prognostic marker in HNSCC.

ELIGIBILITY:
Inclusion Criteria:

* Histological proven squamous cell carcinoma of the pharynx, larynx, oropharynx and hypopharynx
* Curative intent and no prior treatment
* Age >= 18 years
* stage T1-4 N0-N3 M0.
* Informed consent according to local guidelines and national law
* The patient is able (psychological, sociological, geographical and physical) to carry through the treatment and follow-up
* Fertile women must use contraceptive devices (IUD or oral contraceptives)

Exclusion Criteria:

* No serious concurrent medical disease
* No metastasis
* No prior disease that can affect the treatment, evaluation or outcome of current disease
* No pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: head and neck cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Can 18F-FAZA can be used as a prognostic marker in HNSCC? | 1, 5 years

SECONDARY OUTCOMES:
Determine the changes in hypoxia in solid tumours as assessed by 18F-FAZA PET during radiotherapy | Patients will be scanned prior to treatment, every 2 weeks during their treatment and once following radiation

CONTACTS AND LOCATIONS:
Overall Officials: Jens Overgaard, Prof., MD, Principal Investigator — Danish Head and Neck Cancer Group (DAHANCA)
Locations (1):
- Department of Oncology, Aarhus University Hospital, Aarhus, Aarhus, Denmark